CLINICAL TRIAL: NCT03607786
Title: The Effect of Combination of Selective Antegrade Cerebral Perfusion With Retrograde Inferior Vena Caval Perfusion on the Outcomes in Patients Underwent Total Aortic Arch Replacement
Brief Title: Antegrade Cerebral Perfusion and Retrograde Inferior Vena Caval Perfusion for Total Aortic Arch Replacement
Acronym: CARTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Du, M.D, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WCH-2018-24
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Type A Aortic Dissection; Circulatory Arrest; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIVP group (Active Comparator): After total cardiopulmonary bypass was initiated, the patient is cooled slowly to induce moderate hypothermia(28-30℃). The combination of selective antegrade cerebral perfusion and retrograde inferior vena caval perfusion is performed. The antegrade perfusion flow rate was is maintained at 6-12 mL/min/kg.Pump pressure of retrograde perfusion was is maintained at 20-30 mmHg, and blood flow was is maintained at 8-12 mL/min/kg.
  Interventions: Procedure: Retrograde Inferior Vena Caval Perfusion
- ACP group (Active Comparator): After total cardiopulmonary bypass was initiated, the patient is cooled slowly to induce moderate hypothermia(26-28℃). Only select antegrade cerebral perfusion is performed by maintaining the flow rate at 6-12 mL/min/kg.
  Interventions: Procedure: Select antegrade cerebral perfusion

INTERVENTIONS:
Procedure: Retrograde Inferior Vena Caval Perfusion — Retrograde Inferior Vena Caval Perfusion is achieved by tethering the inferior vena cava with a band around the cannula and by clamping the distal end of the inferior vena cava drainage tube, which allowed a pump to drive oxygenated blood into the inferior vena cava. Pump pressure is maintained at 20-30 mmHg, and blood flow is maintained at 8-12 mL/min/kg. The aim of RIVP is to maintain the lower body perfusion during circulation arrest, and reduce the ischemia-associated vital organ injury.
  Other Names: Select antegrade cerebral perfusion
  Arms: RIVP group
Procedure: Select antegrade cerebral perfusion — Antegrade cerebral perfusion is achieved using a 12 F cannula inserted into the brachiocephalic artery or right axillary artery. The antegrade perfusion flow rate is maintained at 6-12 mL/min/kg
  Arms: ACP group

SUMMARY:
This study is designed as a multicenter, randomized, assessor- blinded clinical trial.The primary aim of this trial is to assess whether retrograde inferior venal caval perfusion combined selective antegrade cerebral perfusion(ACP)under mild hypothermia, compared with moderate hypothermia combined with selective ACP alone, improves the outcome for the patients undergoing total aortic arch replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 yr-65yr
2. Patient underwent total aortic arch replacement

Exclusion Criteria:

1. Inability to understand/give informed consent,
2. Participation in another clinical trial that interferes with the primary or secondary outcomes of this trial.
3. Inability to obtain superior and inferior vena caval cannulation due to pericardium adhesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite major complications | up to 12 months
  Newly Postoperative Renal Failure;Surgical Re-exploration；Operative Mortality;Deep Sternal Wound Infection;Stroke/Cerebrovascular Accident;Paraplegia

SECONDARY OUTCOMES:
Respiratory Failure | up to 30 days
Transient Neurological Deficit | up to 30 days
  The occurrence of postoperative agitation, confusion, delirium, obtundation or a transient focal neurologic deficit (resolution within 72 hours) without any evidence of new structural abnormality on computed tomography or magnetic resonance imaging.
Acute Kidney Injury not requiring Dialysis | up to 30 days
  Kidney Disease Improving Global Outcomes (KDIGO) guidelines17
Myocardial Infarction | up to 30 days
Postoperative Prolonged Intubation | up to 30 days
  patients aged 18 years and older who require intubation for more than 24 hours patients aged 18 years and older undergoing isolated CABG who require intubation for more than 24 hours patients aged 18 years and older undergoing isolated CABG who require intubation for more than 24 hours patients aged 18 years and older undergoing isolated CABG who require intubation for more than 24 hours Patients who require intubation for more than 24 hours
Paraparesis | up to 30 days
  Motor weakness in any lower extremity muscle group or unilateral paraplegia (Tarlov score 1-4 or, if present, a score of zero in a single lower extremity)

OTHER OUTCOMES:
The number of volume of blood products transfusion | up to 30 days
  The number of units of packed red blood cells , fresh-frozen plasma, pooled platelets and cryoprecipitate administered was collected from blood bank records
Length of ICU stay | up to 30 days
  The duration of staying ICU postoperatively, time between administrated in ICU after the procedure to discharge from the ICU
Length of postoperative stay | up to 30 days
  the number of days between procedure and discharge, including any time patients spent at hospitals or long-term acute care facilities after transfer from our institution
Gastrointestinal bleed | up to 30 days
  Gastrointestinal bleed is defined as unambiguous clinical or endoscopic evidence of blood in the gastrointestinal tract. Upper gastrointestinal bleeding (or haemorrhage) is that originating proximal to the ligament of Treitz, in practice from the oesophagus, stomach and duodenum. Lower gastrointestinal bleeding is that originating from the small bowel or colon.
Postoperative ascites | up to 30 days
  Accumulation or retention of free fluid in the abdominal peritoneal cavity between the tissues lining the abdomen and abdominal organs. The fluid may be serous, hemorrhagic, or the result of inflammation or tumor metastasis to the peritoneum.
Death | 12 months
  since incident surgery
New onset dialysis (since incident surgery) status | 12 months
  Renal failure requiring dialysis
Stroke | 12 months
  Any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain
Myocardial infarction | 12 months
  Increase in serum cardiac biomarker values (preferably cardiac troponin) with at least one value above the 99th percentile upper reference limit and at least one of the following criteria: symptoms of ischaemia; new or presumed new significant ST segment or T wave ECG changes or new left bundle branch block; development of pathological Q waves on ECG; radiological or echocardiographic evidence of new loss of viable myocardium or new regional wall motion abnormality; identification of an intracoronary thrombus at angiography or autopsy（since incident surgery）

CONTACTS AND LOCATIONS:
Overall Officials: Lei Du, M.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Lin J, Qin Z, Liu X, Xiong J, Wu Z, Guo Y, Kang D, Du L. Retrograde inferior vena caval perfusion for total aortic arch replacement surgery: a randomized pilot study. BMC Cardiovasc Disord. 2021 Apr 20;21(1):193. doi: 10.1186/s12872-021-02002-9. PMID 33879045
- [Derived] Lin J, Tan Z, Yao H, Hu X, Zhang D, Zhao Y, Xiong J, Dou B, Zhu X, Wu Z, Guo Y, Kang D, Du L. Retrograde Inferior Vena caval Perfusion for Total Aortic arch Replacement Surgery (RIVP-TARS): study protocol for a multicenter, randomized controlled trial. Trials. 2019 Apr 24;20(1):232. doi: 10.1186/s13063-019-3319-2. PMID 31014386